CLINICAL TRIAL: NCT03266965
Title: Histaminergic Basis of Central Fatigue in Multiple Sclerosis - A Novel Approach
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kottil W. Rammohan, Professor Of Clinical Neurology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20161186; W81XWH-16-1-0462 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2017-07-04; First posted 2017-08-30 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis
Keywords: Fatigue; Histamine
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Carbidopa; Histidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Histidine Intervention Group (Experimental): A total of 15 subjects will be recruited in batches of 5 until completed 15 subjects in the trial. If a subject withdraws the trial, the study will continue and enrolling subjects until 15 of them complete the trial. The subject composition (MS patient/Normal subject) 4 MS and 1 normal will be tested on a dose of L-Histidine 250 mg plus Lodosyn 50 mg BID for seven days. If there are no safety concerns, the next 5 patients will be recruited 4 MS and 1 normal to test the dose of 500 mg with Lodosyn 50 mg bid for seven days. If there are no safety concerns, then L-histidine 1,000 mg plus Lodosyn (Carbidopa) 50 mg bid will be tested in the next 5 subjects 4 MS and 1 normal for seven days.
  Interventions: Drug: Carbidopa; Dietary Supplement: L-Histidine

INTERVENTIONS:
Drug: Carbidopa — All subjects will receive a fixed dose of 50mg of Lodosyn twice daily.
  Other Names: Lodosyn
Dietary Supplement: L-Histidine — Sequential Dose Escalation of 250mg to 500mg to 1000mg twice daily.

SUMMARY:
The histaminergic system is phylogenetically one of the oldest parts of the nervous system but it is a relatively recent discovery. It is involved with several vegetative functions like sleep, attention and learning, feeding and satiety, working memory, cognition, depression, and most of all arousal and energy

DETAILED DESCRIPTION:
1. Establish in an open label clinical trial the tolerability and safety of various doses of l-histidine and lodosyn that may increase levels of l-histidine and histamine in the serum and cerebrospinal fluid (CSF).
2. Perform pharmacokinetic studies in serum and CSF of study subjects the levels of l-histidine and histamine after treatment with various combination of l-histidine and lodosyn.
3. Preliminary information will also be collected on the effects of this intervention on alleviation of fatigue.

The findings from this study go beyond the effects of histamine on fatigue. If central histamine can be increased by the strategy outlined above, a number of other vegetative hypothalamic functions intricately associated with fatigue including sleep, cognition and satiety need to be examined in MS patients in future studies.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers:

1. Male or female subjects between the ages of 18 and 60 will be eligible.
2. Subjects should be in good physical health without history of chronic illness and should be generally considered healthy.
3. Spouses or caregivers of patients with MS would be encouraged to participate.

Inclusion Criteria for Patients with Multiple Sclerosis (MS):

1. Patients with MS regardless of the disease type, who experience severe fatigue will be eligible to participate.
2. Fatigue Severity Score of >/= 4.0 will qualify as long as all other inclusion / exclusion criteria are met.
3. Established MS by McDonald Criteria - 2010 Revision (24). Relapse Remitting (RR) and progressive forms of MS are eligible
4. Severe fatigue that has lasted greater than 6 months
5. Clinically stable on a current therapy with any Disease Modifying Therapy (DMT)

Exclusion Criteria for Healthy Volunteers:

1. Adults unable to give informed consent due to cognitive impairment or mental disorders.
2. Children below the age of consent
3. Pregnant women
4. Prisoners
5. History of chronic disorders like hypertension, diabetes, hyperlipidemia, depression, hypothyroidism etc. that require chronic treatment
6. Known chronic fatigue syndrome
7. Blood disorders or coagulopathy
8. Chronic allergies or history of asthma.
9. Using antihistamines, bronchodilators or H2 blockers for hyperacidity
10. Using medications for sleep, or known sleep disorders
11. Any medication or condition deemed unsuitable by the PI

Exclusion Criteria for Patients with Multiple Sclerosis (MS):

1. Adults unable to give informed consent due to cognitive impairment or mental disorders.
2. Children below the age of consent
3. Pregnant women
4. Prisoners
5. Systemic disorders known to cause fatigue such as severe anemia, infections, chronic systemic infectious or inflammatory disorders, including known autoimmune disorders.
6. Chronic fatigue syndrome
7. Hypothyroidism
8. Systemic malignancy
9. Undergoing chemotherapy
10. Depression
11. Sleep disorders including narcolepsy, excessive day-time sleep.
12. History of substance abuse
13. Excessive consumption of coffee or over-the-counter stimulants
14. Concomitant medications of amantadine, methylphenidate, amphetamines, pemoline, barbiturates, tizanidine, Monoamine oxidase inhibitor (MAO) inhibitors, benzodiazepines, barbiturates, tricyclic antidepressants, antihistamines, H2 blockers for gastro-esophageal reflux disease (GERD), selective serotonin reuptake inhibitors (SSRIs) and any other medication that in the opinion of the PI should be excluded.
15. Patients who were using modafinil for treatment of fatigues prior to the study may participate but will be required to undergo a washout of 2 weeks prior to entry into the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events experienced by participants. | 30 days
  All adverse and serious adverse events reported during the study will be analyzed and tabulated. No quantitative statistical analysis will be performed. The primary goal of this study is to establish that this intervention is safe and possibly effective.

SECONDARY OUTCOMES:
Change extent of fatigue. | Screening(0 day), baseline(15 days) and final visit(30 days)
  At the conclusion of the study, each individual would have completed a screening and baseline visit without any intervention and two weekly visits during intervention with the study medications. The two evaluations off drug will be compared to the two evaluations on drug. A drop of the Fatigue Severity Scale (FSS) score by 1 point or more will be considered a response. Once the information is converted into a binary function of response / no response, the data is amenable to conditional logistic regression analysis.
Change in Quality of life. | Screening(0 day), baseline(15 days) and final visit(30 days)
  Multiple Sclerosis Quality of Life (MSQOL) scales will be used to measure the change in Quality of Life. Based on the scale, there will be a 0 to 100 with a higher score indicating a higher quality of life.
Change of fatigue impact scale. | Screening(0 day), baseline(15 days) and final visit(30 days)
  Modified Fatigue Impact Scale (MFIS) scale will be used to evaluate the physical, cognitive and psychosocial scores. The score ranges from 0 to 84 with a lower score, lower side effects of fatigue.
Change of visual pain. | Screening(0 day), baseline(15 days) and final visit(30 days)
  Visual analogue scale to evaluate the pain by using a numerical scale for 0 to 10 with a lower score, less visual pain.
Change of daytime sleepiness. | Screening(0 day), baseline(15 days) and final visit(30 days)
  Epworth sleep scale to rate the probability of falling asleep during daytime on a scale of 0 to 24 with a lower score the lower the symptoms of sleepness.
Change of hunger sensitivity. | Screening(0 day), baseline(15 days) and final visit(30 days)
  Hunger Satiety Scale to determine the extent of hunger and fullness by using a 1 to 10 score range with a higher score indicating a higher hunger sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Kottil Rammohan, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No